CLINICAL TRIAL: NCT03433872
Title: Professional Development Tools to Improve the Quality of Infant and Toddler Care
Acronym: Q-CCIIT PD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mathematica Policy Research, Inc. (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency); University of Oklahoma (Other); Zero to Three (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 50192
Record Dates: First submitted 2018-01-23; First posted 2018-02-15 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Early Childhood Professional Development
Keywords: Infant-toddler care; Early child development; Professional development

STUDY DESIGN:
Intervention Model Description: The goal of the field test is to evaluate use of the We Grow Together system by typical early childhood professionals working in a variety of care settings serving infants and toddlers. The field test will take place in 8 to 12 geographic areas across the country. This study will include only centers and FCC settings that already have local PD providers-the investigators will exclude ECE settings without established PD providers. The field test will include a purposive sample of 175 center-based classrooms (approximately half will be affiliated with Early Head Start [EHS], and half will be community-based child care programs). The field test sample will also include 125 FCCs, including those operating under EHS and in community-based settings.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Caregivers (Other): "Caregiver" refers to teachers and child care providers in infant and toddler classrooms in center-based or FCC settings. All caregivers in the study will be assigned to the intervention. The PD providers supporting these caregivers will be trained in the We Grow Together: The Q-CCIIT Professional Development System.
  Interventions: Other: We Grow Together: The Q-CCIIT Professional Development System

INTERVENTIONS:
Other: We Grow Together: The Q-CCIIT Professional Development System — We Grow Together is designed to strengthen high quality caregiver interactions with infants and toddlers. The starting point for the We Grow Together study is assessment of a caregiver's interactions with infants and toddlers in the caregiver's ECE setting, using the Q-CCIIT observational measure. Data from the Q CCIIT observations highlight areas for growth in the caregiver's practices and will inform a PD goal-setting process, with the help of a PD Provider. An array of We Grow Together materials targeting practices assessed by the Q-CCIIT measure and informed by professional development and behavior change research are organized into modules, and delivered on an interactive website. Over the course of a program year, each caregiver in the study will work with a PD provider who is trained in guiding caregivers through the use of We Grow Together materials.

SUMMARY:
Mathematica Policy Research, funded by OPRE, ACF, DHHS, will conduct a field test of We Grow Together: The Q-CCIIT Professional Development System. These professional development (PD) tools and the interactive website featuring the materials were developed to promote high-quality caregiver-child interactions in non-parental care settings serving infants and toddlers. This field test aims to: (1) examine changes in caregiver practice that the investigators expect to be associated with use of the We Grow Together system, and (2) examine implementation of We Grow Together. As a secondary goal, the investigators will further evaluate the psychometrics of the Q-CCIIT observational measure of interaction quality.

Collecting data from field test participants will occur from fall 2018 through spring 2019. First, the investigators plan to collect a background survey with caregivers and PD providers in fall 2018. Second, in fall 2018 and spring 2019 the investigators plan two rounds of classroom observations using the Q-CCIIT measure and classroom rosters. Third, the investigators plan to collect data on the use and implementation of We Grow Together through the interactive website from fall 2018 through spring 2019. Finally, the investigators plan to conduct a feedback survey with caregivers and PD providers in spring 2019.

DETAILED DESCRIPTION:
The We Grow Together intervention is designed to help caregivers understand how caregiver interactions with children support the children's development to strengthen high quality caregiver interactions with infants and toddlers. The starting point for the We Grow Together process is assessment of a caregiver's interactions with infants and toddlers in early childhood care and education (ECE) settings, using the Quality of Caregiver-Child Interactions with Infants and Toddlers (Q-CCIIT) observational measure. Data from the Q CCIIT observations highlight areas for growth in the caregiver's practices and inform a PD goal-setting process, with the support of a PD Provider.

The investigators have developed an array of We Grow Together materials targeting principles and practices assessed by the Q-CCIIT measure, organized into modules, and delivered on an interactive website. Over the course of a program year, each caregiver in the study will work with a PD provider who is trained in guiding caregivers through the use of We Grow Together materials.

As part of the We Grow Together intervention, all PD providers will receive training in using We Grow Together to support caregivers' understanding and practices. PD providers' training will focus on understanding the caregiving principles, relationship skills, adult learning principles, and coaching strategies that facilitate use of We Grow Together and promote growth of caregivers' knowledge and skills. PD providers will also have access to a set of PD provider materials to support implementation of We Grow Together. These materials support the ongoing relationship-based PD between the PD Provider and caregiver.

The purpose of information collected under the current request is to examine the implementation and the outcomes associated with use of We Grow Together. The goals of the field test will be to: (1) implement We Grow Together for five months in a variety of settings, (2) collect information on the implementation of We Grow Together, and (3) collect information on care practices the investigators hypothesize are associated with use of We Grow Together. The investigators propose the following data collection activities, to be carried out in fall 2018 through spring 2019:

* An ECE setting eligibility screening will determine if a setting is eligible and if family child care (FCC) and center directors and individual personnel are willing to participate in the field test.
* A background survey, completed by all caregivers and PD providers
* Observations of caregiver interactions by the investigators using the Q-CCIIT measure, to assess the quality of care provided by participating caregivers.
* A classroom information roster, completed by caregivers at the time of the observation, about the composition and activities within care settings.
* Web-user pop-up questions for caregivers and PD providers, collected monthly at website login.
* A feedback survey, completed by caregivers and PD providers.
* A PD provider training survey.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the study caregivers and PD providers in center-based and FCC ECE settings must meet the following criteria:

1. Operate within one of the selected geographical areas.
2. Caregivers must have a current PD provider with whom the caregiver works one-on-one with at least once a month.
3. Serve children between the ages of birth to 36 months.
4. Written knowledge of English.
5. Caregivers and PD providers must agree to participate in the We Grow Together professional development system for approximately 5 months.

Exclusion Criteria:

* Does not meet the inclusion criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 475 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Quality of Caregiver Child Interaction with Infant and Toddlers (Q-CCIIT) | 2-3 hours
  Observational measure
Beliefs about Infant-Toddler Development | Up to 3 months
  Study developed survey of knowledge and beliefs about child development
Beliefs about Infant-Toddler Caregiving | Up to 3 months
  Study developed survey of beliefs about quality care for infants and toddlers
Self-reported beliefs about PD | Up to 3 months
  Study developed survey of professional development
Use of website PD tools | Up to 5 months
  Website analytics (metadata)
Satisfaction with We Grow Together professional development system | Up to 3 months
  Study developed survey of professional development
Use of PD strategies | Up to 3 months
  Study developed survey of professional development